CLINICAL TRIAL: NCT00311545
Title: A Phase II Study of CNTO 328, A Monoclonal Antibody Against Interleukin-6 (IL-6), In Patients With Advanced or Metastatic Renal Cell Cancer
Brief Title: S0351, CNTO 328 in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawal of support for drug supply
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462096; S0351 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; stage III renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CNTO 328 (Experimental): CNTO 328, anti-IL-6 monoclonal antibody; 6 mg/kg, IV, q 2wks x 12 cycles (1 cycle = 2 wks)
  Interventions: Biological: CNTO 328

INTERVENTIONS:
Biological: CNTO 328 — Anti-IL-6 chimeric monoclonal antibody
  Other Names: Siltuximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as CNTO 328, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well CNTO 328 works in treating patients with unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the probability of response (confirmed complete and partial responses) in patients with unresectable or metastatic renal cell cancer treated with CNTO 328.

Secondary

* Assess the 6-month progression-free survival probability and median overall survival in these patients.
* Evaluate the qualitative and quantitative toxicities of this treatment.
* Investigate, in a preliminary manner, the association of tumor response with potential markers of anti-interleukin-6 activity.

OUTLINE: This is a multicenter study.

Patients receive CNTO 328 IV over 2 hours on day 1. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete or partial response after 6 courses of therapy may receive an additional 6 courses.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or unresectable primary renal cell carcinoma
* Measurable disease

  * Soft tissue disease within a prior radiation field may be considered measurable disease provided all of the following are true:

    * Patient also has measurable disease outside of the irradiated field
    * Disease within the irradiated field has progressed since prior radiotherapy
    * Radiotherapy was completed more than 2 months ago
* Ineligible for high-dose interleukin-2
* No treated or untreated brain metastases

  * No history of brain metastases
  * Patients with clinical evidence of brain metastases must have brain CT scan or MRI negative for metastatic disease within 56 days prior to study entry

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance ≥ 40 mL/min
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* SGOT ≤ 3 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No more than 2 of the following:

  * Zubrod PS 2
  * Lactate dehydrogenase > 1.5 times ULN
  * Hemoglobin < lower limit of normal
  * Calcium > 10 mg/dL
  * Absence of prior nephrectomy
* No uncontrolled intercurrent illness, including any of the following:

  * Uncontrolled diabetes mellitus
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No HIV positivity
* No other prior malignancy, excluding the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer for which the patient is currently in complete remission
  * Any other cancer for which the patient has been disease free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 28 days since prior tumor resection and recovered
* No prior immunotherapy or chemotherapy regimens with interferon (IFN) and/or interleukin-2 (IL-2) or the combination of IFN/IL-2
* No prior cytotoxic chemotherapy for renal cell cancer
* No prior murine or chimeric proteins or human/murine recombination products (i.e., other chimeric monoclonal antibodies)
* No concurrent radiotherapy or systemic therapy for renal cell cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek K. Pinski, MD, Study Chair — University of Southern California; Philip C. Mack, Ph.D., Study Chair — UC Davis Cancer Center